CLINICAL TRIAL: NCT04986085
Title: Nutritional Status of Patients With Gastroenteropancreatic Neuroendocrine Tumors in Spain: NUTRIGETNE
Brief Title: Nutrition in Gastroenteropancreatic Neuroendocrine Tumor
Acronym: NUTRIGETNE
Status: Completed | Type: Observational
Sponsor: Grupo Espanol de Tumores Neuroendocrinos (Other)
Responsible Party: Sponsor
Other Study IDs: GETNE-S2109
Record Dates: First submitted 2021-03-22; First posted 2021-08-02 (Actual); Results first posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Gastroenteropancreatic Neuroendocrine Tumor
Keywords: GEP NET; Neuroendocrine tumor; Nutritional status
MeSH Terms: conditions — Gastro-enteropancreatic neuroendocrine tumor; Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GEP NET: GEP NET patients in Spain

SUMMARY:
It is well known that the prevalence of malnutrition or risk of malnutrition in cancer patients is high, as well as its impact on different parameters such as hospitalization, survival or response to certain treatments. In patients with gastroenteropancreatic (GEP) neuroendocrine tumors (NET), due to their heterogeneity and longer survival, it is expected that the prevalence of malnutrition is probably underdiagnosed, as well as the existence of a negative impact on different parameters (quality of life, survival). So far, the studies carried out on nutrition and NET are very scarce and none has been carried out so far in Spain.

Before being able to carry out nutritional intervention studies on these patients, it is necessary to know the reality of the nutritional status of patients with NETs in Spain. The main motivation for the NUTRIGETNE study is to evaluate the epidemiological status of nutrition in NETs in the spanish population. In addition to know the epidemiological picture, it is intended to study the nutritional status from different points of view: analytical, clinical, anthropometric, etc. Besides, the study of nutritional status will allow us to closely monitor the patients who have a higher risk of malnutrition and to propose early interventions for those, as well as the impact of their nutritional status on different parameters: survival, hospitalization, quality of life or responses to the treatments.

NUTRIGETNE is a cross-sectional, open and multicenter study in which the nutritional status of patients with GEP NET in Spain will be evaluated.

DETAILED DESCRIPTION:
NUTRIGETNE is a cross-sectional, open and multicenter study in which the nutritional status of patients with GEP NET in Spain will be evaluated. It is planned to include 400 GEP NET patients. Patients will be included consecutively when visiting the corresponding health centers for outpatient visits or hospitalization.

The study comprises 3 stages with a total duration of 10 to 40 days for the participation of each subject in the study:

Screening visit, First day (day 0): The initial screening will take place on the first day the patient visits the hospital. The inclusion and exclusion criteria will be reviewed to assess the eligibility of the patient. The implications of the study will be explained to the patient and the informed consent will be signed.

Visit for assessment of nutritional status (days 0-10): taking a medical history, complete physical examination including anthropometry, bioelectrical impedance (BIA) and dynamometry, as well as laboratory analysis. The evaluation of the nutritional status will be carried out by a registered nutritionist, specialized nurse or specialist doctor (variable depending on the characteristics of the center).

Data collection (day 10-40): collection of analytical, anthropometric, BIA, dynamometry and clinical results and introduction into the electronic case report form (eCRF).

After the end of recruitment and database lock, all data will be subsequently analyzed and presented when applicable through study reports and scientific communications.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with a gastroenteropancreatic neuroendocrine tumor by histopathological study.
* Legally capable patients ≥ 18 and ≤ 80 years of age.
* Patients who have signed the informed consent for this study as specified in section 10.3.
* Patients in active treatment: active treatment is considered to be those patients in an advanced stage and in any type of medical treatment (somatostatin analogues, molecular therapies, chemotherapy, radionuclides...), or locoregional therapies.

Note: Decision was taken to treat the patient with an specific treatment prior and independently of patient inclusion in this non interventional study.

Exclusion Criteria:

* Patients <18 or > 80 years of age.
* Female patients that are currently pregnant.
* Patients with a gastroenteropancreatic neuroendocrine tumor lacking an histopathological diagnosis.
* Patients in palliative treatment or terminal stage.
* Patients who have not signed the informed consent or any situation or condition that compromises the giving of patient voluntary informed consent.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with gastroenteropancreatic neuroendocrine tumors diagnosed histologically that are on active treatment for the disease in Spain
Sampling Method: Probability Sample
Enrollment: 399 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: María Isabel del Olmo García, M.D. Ph.D., Principal Investigator — Hospital Universitario La Fe; María Argente Pla, M.D. Ph.D., Principal Investigator — Hospital Universitario La Fe
Locations (16):
- Spain (16):
  - Hospital Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Universitario Vall d´Hebron, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario de Cabueñes, Gijón
  - Hospital Universitario Dr. Josep Trueta, Girona
  - Hospital Universitario la Princesa, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario la Paz, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela
  - Hospital Universitari i Poliècnic la Fe, Valencia
  - Institut Valencià d'Oncologia (IVO), Valencia
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GEP NET
Started | 399
Completed | 399
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Full dataset
Arm/Group | GEP NET
Number analyzed (Participants) | 399
Age, Continuous [Median (Full Range); unit: years] | 62 [22 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 171
  Male | 228
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 380
  Hispanic or latino | 13
  African | 6
Region of Enrollment [Number; unit: participants]
  Spain | 399
Eastern Cooperative Oncology Group performance status (ECOG-PS) [Count of Participants; unit: Participants] — The ECOG PS score describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.).
  The score ranges from 0 (Fully active, able to carry on all pre-disease performance without restriction) to 5 (dead)
  Participants
    Score 0 | 213
    Score 1 | 125
    Score ≥ 2 | 20
    Score Unknown | 41
Tumor grade; World Health Organization (WHO) [Count of Participants; unit: Participants] — The pathologist gives the NET a grade from 1 to 3. A lower number means the tumour is a lower grade. The factors used to determine the grade for NETs include: how often the cells of the tumour are dividing (measured as mitotic count and Ki-67 labelling index). Higher grade indicates a less differentiated tumor with more aggressive behaviour
  Participants
    Grade 1 | 147
    Grade 2 | 197
    Grade 3 | 50
    Unknown | 5
Tumor Differentiation [Count of Participants; unit: Participants] — Well-differentiated neuroendocrine tumors (NETs): The cells resemble and behave like normal cells and tend to grow slowly. Most Grade 1 and Grade 2 NETs are this type. Poorly differentiated neuroendocrine carcinomas (NEC): These cells look abnormal and don't resemble or behave like normal cells. They tend to grow fast.
  Participants
    Tumors (NET) | 361
    Carcinomas (NEC) | 28
    Unknown | 10
Functionality [Count of Participants; unit: Participants] — Some tumours (functioning tumours) may cause abnormally large amounts of hormones to be released into the bloodstream. This can cause symptoms such as diarrhoea, flushing, cramps, wheezing, low blood sugar (hypoglycaemia), changes in blood pressure and heart problems
  Participants
    Functioning | 98
    Not functioning | 295
    Unknown | 6
Primary tumor location [Count of Participants; unit: Participants] — Gastroenteropancreatic neuroendocrine neoplasms (GEP-NENs) are epithelial neoplasms with neuroendocrine differentiation that occur inside the gastrointestinal (GI) tract and the pancreas. Some tumors may be diagnosed by the presence of metastasis or appearance of symptoms in functioning tumors, while primary tumor remains undetermined, unknown origin.
  Here we report the primary tumor locations
  Participants
    Small intestine | 177
    Pancreas | 167
    Colorectal | 18
    Gastric | 10
    Other / Unknown | 27
Metastasis at inclusion [Count of Participants; unit: Participants] — The metastatic process involves tumor cell invasion of distant organs to the primary tumor site. Presence of metastasis may correlate with worse prognosis in most cases.
  Here we report the number of metastatic locations
  Participants
    0 | 15
    1 | 227
    ≥ 2 | 157
Most common sites of metastasis [Count of Participants; unit: Participants] — Here we report the number of patients who hace metastasis in the most common organs / locations
  Participants
    Liver: Metastasis present | 332
    Liver: No metastasis | 67
    Lymph nodes: Metastasis present | 86
    Lymph nodes: No metastasis | 313
    Peritoneum: Metastasis present | 55
    Peritoneum: No metastasis | 344
    Lung: Metastasis present | 28
    Lung: No metastasis | 371
Previous lines of treatment [Count of Participants; unit: Participants] — Here we report the number of previous systemic treatments received by the patients before the inclusion in the NUTRIGETNE study.
  Participants
    1 | 217
    2 | 92
    ≥ 2 | 90
Type of previous lines [Count of Participants; unit: Participants] — Here we report the type of previous systemic treatments received by the patients before their inclusion in the NUTRIGETNE study.
  Participants
    Somatostatin analogs (SSA): Received this previous treatment | 342
    Somatostatin analogs (SSA): Not received this previous treatment | 57
    Peptide receptor radiotherapy (PRRT): Received this previous treatment | 109
    Peptide receptor radiotherapy (PRRT): Not received this previous treatment | 290
    Targeted kinase inhibitors: Received this previous treatment | 108
    Targeted kinase inhibitors: Not received this previous treatment | 291
    Chemotherapy: Received this previous treatment | 80
    Chemotherapy: Not received this previous treatment | 319
    Clinical trial: Received this previous treatment | 42
    Clinical trial: Not received this previous treatment | 357
    TACE or locoregional therapy: Received this previous treatment | 11
    TACE or locoregional therapy: Not received this previous treatment | 388
    Immunotherapy: Received this previous treatment | 7
    Immunotherapy: Not received this previous treatment | 392
    Others: Received this previous treatment | 6
    Others: Not received this previous treatment | 393

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Malnutrition in GEP NET
Description: Percentage of GEP NET patients suffering from malnutrition in Spain according to the Global Leadership Initiative on Malnutrition (GLIM), which was convened by several of the major global clinical nutrition societies. Malnutrition diagnosis is based on three phenotypic criteria (non-volitional weight loss, low body mass index, and reduced muscle mass) and two etiologic criteria (reduced food intake or assimilation, and inflammation or disease burden). Patients having one or more phenotypic and etiologic criteria are considered malnourished.
Time Frame: Throughout the study period. Nutritional status will be reported at a single timepoint for each patient (between 1-10 days after informed consent signature)
Measure: Count of Participants; unit: Participants
Arm/Group | GEP NET
Number analyzed (Participants) | 399
Participants
  Malnutrition (GLIM criteria) | 247
  No malnutrition | 152

2. Primary Outcome: Risk of Malnutrition in GEP NET
Description: Percentage of GEP NET patients at risk of suffering from malnutrition in Spain according to Malnutrition Universal Screening Tool (MUST). Three independent criteria are used by MUST to determine the overall risk for malnutrition: current weight status using BMI, unintentional weight loss, and acute disease effect.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GEP NET
Number analyzed (Participants) | 399
Participants
  Low risk | 264
  Intermediate risk | 67
  High risk | 56
  Missing | 12

3. Secondary Outcome: Body Mass Index
Description: Body mass index (BMI) is defined as a a measure of body fat based on height and weight that applies to adult men and women
Time Frame: as for outcome 1
Population: The endpoint is reported in overall population and in subgroups. according to their sex and malnutrition status.
  The analyzed patient number in each subgroup might be inferior to the full sample size as some patients may have missing BMI , or unknown GLIM malnutrition status.
Measure: Count of Participants; unit: Participants
Arm/Group | GEP NET
Number analyzed (Participants) | 399
Participants
  Male: number analyzed (Participants) | 228
  Male: Underweight (BMI < 18.5) | 6
  Male: Normal (BMI 18.5 - 25) | 96
  Male: Overweight (BMI 25 - 30) | 95
  Male: Obese (BMI >= 30) | 31
  Female: number analyzed (Participants) | 171
  Female: Underweight (BMI < 18.5) | 17
  Female: Normal (BMI 18.5 - 25) | 89
  Female: Overweight (BMI 25 - 30) | 53
  Female: Obese (BMI >= 30) | 12
  Malnutrition (GLIM): number analyzed (Participants) | 247
  Malnutrition (GLIM): Underweight (BMI < 18.5) | 23
  Malnutrition (GLIM): Normal (BMI 18.5 - 25) | 116
  Malnutrition (GLIM): Overweight (BMI 25 - 30) | 80
  Malnutrition (GLIM): Obese (BMI >= 30) | 28
  No malnutrition (GLIM): number analyzed (Participants) | 151
  No malnutrition (GLIM): Underweight (BMI < 18.5) | 0
  No malnutrition (GLIM): Normal (BMI 18.5 - 25) | 68
  No malnutrition (GLIM): Overweight (BMI 25 - 30) | 68
  No malnutrition (GLIM): Obese (BMI >= 30) | 15
  Overall: Underweight (BMI < 18.5) | 23
  Overall: Normal (BMI 18.5 - 25) | 185
  Overall: Overweight (BMI 25 - 30) | 148
  Overall: Obese (BMI >= 30) | 43

4. Secondary Outcome: Body Fat
Description: Body fat mass calculated by bioimpedance
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Median (Full Range); unit: Kg
Arm/Group | GEP NET
Number analyzed (Participants) | 399
Kg
  Male: number analyzed (Participants) | 210
  Male | 58.2 [18.4 to 84.5]
  Female: number analyzed (Participants) | 171
  Female | 41.5 [8.7 to 73.5]
  Malnutrition (GLIM): number analyzed (Participants) | 247
  Malnutrition (GLIM) | 47.0 [8.7 to 77.4]
  No Malnutrition (GLIM): number analyzed (Participants) | 151
  No Malnutrition (GLIM) | 57.3 [36.7 to 84.5]
  Overall | 51.4 [8.7 to 84.5]

5. Secondary Outcome: Phase Angle
Description: Body muscle mass calculated by bioimpedance and measured by Phase Angle. Here we report the phase angle, a marker of muscle mass and function, measured in degrees. Higher degrees of phase angle indicates greater cell integrity and function, reflecting healthier and more robust muscles.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Median (Full Range); unit: degrees
Arm/Group | GEP NET
Number analyzed (Participants) | 399
degrees
  Male: number analyzed (Participants) | 228
  Male | 5.5 [1.8 to 9.0]
  Female: number analyzed (Participants) | 171
  Female | 4.8 [3.0 to 11.0]
  Malnutrition (GLIM): number analyzed (Participants) | 247
  Malnutrition (GLIM) | 5.0 [2.2 to 11.0]
  No malnutrition (GLIM): number analyzed (Participants) | 151
  No malnutrition (GLIM) | 5.6 [1.8 to 9.0]
  Overall | 5.1 [1.8 to 11.0]

6. Secondary Outcome: Nutritional Risk Screening (NRS) Rates
Description: Scale to evaluate the malnutrition in adult patients. It is based in the assessment of BMI, weight loss in the last 3-6 months and acute disease effects. The score ranges from 0 (low malnutrition risk to 6 (high malnutrition risk).
Time Frame: as for outcome 1
Population: The endpoint is reported in overall population and in subgroups. according to the malnutrition status. The analyzed patient number in each subgroup might be inferior to the full sample size as some patients may have missing BMI , or unknown GLIM malnutrition status.
Measure: Median (95% Confidence Interval); unit: Score
Arm/Group | GEP NET
Number analyzed (Participants) | 399
Score
  Malnutrition (GLIM): number analyzed (Participants) | 247
  Malnutrition (GLIM) | 1.5 [0 to 5]
  No malnutrition (GLIM): number analyzed (Participants) | 151
  No malnutrition (GLIM) | 0 [0 to 4]
  Overall | 1 [0 to 2]

7. Secondary Outcome: Subjective Global Assessment (SGA) Rates
Description: Score to measure risk malnutrition in adult patients based on patient history and physical examination alone. The score has 3 levels: A (low malnutrition risk) to C (high malnutrition risk)
Time Frame: as for outcome 1
Population: The endpoint is reported in overall population and in subgroups. according to the malnutrition status
Measure: Count of Participants; unit: Participants
Arm/Group | GEP NET
Number analyzed (Participants) | 399
Participants
  Malnutrition (GLIM): number analyzed (Participants) | 245
  Malnutrition (GLIM): Good nutritional status | 144
  Malnutrition (GLIM): Moderate malnutrition or risk of malnutrition | 79
  Malnutrition (GLIM): Severe malnutrition | 22
  Malnutrition (GLIM): Missing data | 0
  No malnutrition (GLIM): number analyzed (Participants) | 149
  No malnutrition (GLIM): Good nutritional status | 140
  No malnutrition (GLIM): Moderate malnutrition or risk of malnutrition | 8
  No malnutrition (GLIM): Severe malnutrition | 1
  No malnutrition (GLIM): Missing data | 0
  Overall: Good nutritional status | 285
  Overall: Moderate malnutrition or risk of malnutrition | 87
  Overall: Severe malnutrition | 23
  Overall: Missing data | 4

ADVERSE EVENTS:
Time Frame: Deaths and Adverse Events were not assessed. Safety was not within the scope of this observational study and was not assessed. The study is a single point visit. There is no prospective data collected.
Description: Not assessed
Arm/Group | GEP NET
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-12): https://cdn.clinicaltrials.gov/large-docs/85/NCT04986085/Prot_SAP_000.pdf